CLINICAL TRIAL: NCT00543608
Title: Randomized, Double-Blind, Multicenter Study to Evaluate Efficacy and Safety of Intravenous Iclaprim Versus Vancomycin in the Treatment of Hospital-Acquired, Ventilator-Associated, or Health-Care-Associated Pneumonia Suspected or Confirmed to be Due to Gram-Positive Pathogens
Brief Title: Clinical Efficacy of Intravenous Iclaprim Versus Vancomycin in the Treatment of Hospital-Acquired, Ventilator-Associated, or Health-Care-Associated Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated due to financial resource limitations
Sponsor: Arpida AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICLA-20-PNE1
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Hospital-Acquired Pneumonia; Ventilator-Associated Pneumonia; Health-Care-Associated Pneumonia
Keywords: pneumonia; nosocomial pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Pneumonia | interventions — iclaprim; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Dose 1 iclaprim
  Interventions: Drug: iclaprim
- 2 (Experimental): Dose 2 iclaprim
  Interventions: Drug: iclaprim
- 3 (Active Comparator): vancomycin
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: iclaprim
  Arms: 1; 2
Drug: vancomycin
  Arms: 3

SUMMARY:
The purpose of this study is to compare the clinical cure rates of two dosing regimens of iclaprim with vancomycin (every 12 hours [q12h]) in the treatment of patients with hospital-acquired pneumonia (HAP), ventilator-associated pneumonia (VAP), or health-care-associated pneumonia (HCAP) suspected or confirmed to be due to Gram-positive pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed acute bacterial pneumonia due to Gram-positive pathogens in one of the following subgroups:

  * hospital-acquired pneumonia (HAP), i.e., pneumonia that occurs 48 hours or more after admission, which was not incubating at the time of admission; or
  * ventilator-associated pneumonia (VAP), i.e., pneumonia that arises more than 48 hours after endotracheal intubation; or
  * health-care-associated pneumonia (HCAP), i.e., pneumonia diagnosed within 48 hours of hospital admission, in a patient who fulfills at least one of the following criteria:

    1. hospitalization for at least two days within 90 days of the current infection,
    2. residence in a nursing home or long-term care facility,
    3. recipient of intravenous antibiotic therapy, chemotherapy, or wound care within 30 days of the current infection

Exclusion Criteria:

* Acute Physiology and Chronic Health Enquiry (APACHE) II score < 8 or ≥ 25.
* Pneumonia not requiring empiric or targeted treatment effective against Gram-positive pathogens.
* Pulmonary infection due to Gram-positive organisms known to be resistant to either study medication prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-04 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Clinical cure rate - comparison of the two iclaprim dosing regimens versus vancomycin | at test of cure (TOC) visit
Efficacy: Iclaprim clinical cure rates | at TOC and end of therapy (EOT)
Safety

CONTACTS AND LOCATIONS:
Overall Officials: David Willms, MD, Principal Investigator — Sharp HealthCare